CLINICAL TRIAL: NCT01750866
Title: Efficacy and Toxicity of Cabazitaxel in Men 75 Years of Age or Older With Castration-Resistant Prostate Cancer With Progression After Treatment With Docetaxel
Brief Title: Cabazitaxel in Men 75 Years of Age or Older With Castration-Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3811; NCI-2012-02993 (Other: NCI/CTRP)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Castrate-resistant Metastatic Prostate Cancer
Keywords: Prostrate Cancer; Castrate-resistant metastatic prostate cancer; Cabazitaxel
MeSH Terms: interventions — cabazitaxel; XRP6258; Prednisone; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental): Cabazitaxel 25 mg/m2 will be administered by intravenous infusion over 1 hour on Day 1 of every 21-day cycle. Treatment will continue until disease progression, intolerable side effects, or a maximum of 10 cycles of therapy.
  Interventions: Drug: Cabazitaxel; Drug: Prednisone; Drug: Granulocyte colony-stimulating factor (G-CSF)

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel 25 mg/m2 will be administered by intravenous infusion over 1 hour on Day 1 of every 21-day cycle.
  Other Names: taxoid XRP6258; Jevtana; RPR-116258A; XRP6258
Drug: Prednisone — Prednisone 10 mg on Day 1 of the first cycle and continue taking 10 mg po daily for the entire cycle.
Drug: Granulocyte colony-stimulating factor (G-CSF) — Granulocyte colony stimulating factor (Neulasta 6 mg sc) with each cycle, starting with the first cycle, to minimize the risk of complications from neutropenia.

SUMMARY:
Cabazitaxel is already approved by the Food and Drug Administration (FDA) for use in patients with advanced prostrate cancer, following docetaxel therapy. The purpose of this study is to better understand the response and toxicity of cabazitaxel of elderly men (age 75 years and older) with advanced prostate cancer who have progressed during or after treatment with docetaxel. All patients on this study will receive cabazitaxel by intravenous (through a vein) infusion plus prednisone by mouth twice daily, and following the chemotherapy infusions, an injection of a granulocyte colony-stimulating factor (G-CSF). G-CSF will help the body produce more white blood cells, which should help decrease the risk of getting an infection while being treated with cabazitaxel.

DETAILED DESCRIPTION:
This is a single arm, open label, phase II trial of cabazitaxel every 3 weeks in patients who are ≥ 75 years of age with castration-resistant, metastatic prostate cancer who have progressed during or after docetaxel.

Primary objective:

-The primary objective is to determine the efficacy of cabazitaxel in men 75 years of age or older with castration-resistant, metastatic prostate cancer who have progressed during of following treatment with docetaxel.

Secondary objectives:

* To characterize the safety and tolerability of cabazitaxel in patients ≥ 75 years of age
* To determine the PSA response
* To determine the effect of cabazitaxel on functional status using geriatric assessments

Exploratory objectives:

* Determine the effect of therapy with cabazitaxel on the number of circulating tumor cells (CTC)
* To measure the effects of cabazitaxel on apoptosis in CTCs from patients ≥ 75 years of age using H2AX and M30 as biomarkers.
* To determine the relationship between geriatric-focused assessment of comorbidity and functional ability and toxicity and response.

Patients will receive cabazitaxel 25 mg/m2 every 3 weeks with 10 mg prednisone daily until progression, intolerance of therapy, or withdrawal of consent. Patients will receive granulocyte colony stimulating factor (Neulasta 6 mg sc) with each cycle, starting with the first cycle, to minimize the risk of complications from neutropenia. Patients will be followed for 28 days after discontinuation of therapy or death, whichever occurs first. Patients with serious adverse events at the time of removal from the trial will be followed until the toxicities resolve or are deemed irreversible by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, castrate-resistant metastatic prostate cancer without neuroendocrine differentiation or small cell histology
* Age ≥ 75 years of age
* Progressive disease despite:
* Previous therapy with docetaxel
* Progressive disease for study enrollment is defined by either:
* PSA criteria according to the Prostate Cancer Clinical Trials Working Group (PCWG2) criteria with a minimum of three rising PSA levels with an interval of ≥ 1 week between each determination and a PSA at the screening visit of ≥ 2 ng/ml
* Radiographic progression in soft tissue according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria
* Appearance of two or more lesions on a bone
* Previous treatment with abiraterone acetate or enzalutamide is allowed, but last dose must be at least 14 days prior to enrollment in this trial.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Ongoing androgen deprivation with a serum testosterone < 50 ng/dL
* A score of 8-14 on the Mini Nutritional Assessment (MNA) (normal nutritional status or at risk of malnutrition). MNA in Appendix 4 and available at www.mna-elderly.com.
* Patients must have the following laboratory values:
* Hematologic:
* Absolute Neutrophil Count (ANC) >/=1.5x109/L
* Hemoglobin (Hgb) >/=9 g/dl
* Platelets (plt) >/=100x109/L
* Biochemistry :
* Potassium within normal limits or correctable with supplements
* Total calcium (corrected for serum albumin) and phosphorus within normal limits Liver and Kidney Functions
* AST (aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT)and ALT (alanine aminotransferase/glutamic pyruvic transaminase/GPT) ≤ 1.5 x Upper Limit of Normal (ULN)
* Serum bilirubin </= 1 x ULN
* Serum creatinine </= 1.5 x ULN. If creatinine is 1.0 to 1.5 x ULN, creatinine clearance will be calculated according to the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula and only patients with a creatinine clearance > 60 mL/min will be included.
* Life expectancy of ≥ 6 months
* No concomitant anticancer or investigational drug or participation in an investigational trial within 30 days of starting treatment with cabazitaxel. Treatment with nitrosoureas, mitomycin, or monoclonal antibodies, such as trastuzumab, must be ≥ 6 weeks
* Male participants with partners who are of child bearing potential must agree to use double barrier method of birth control 28 days prior to study entry, during the study and for 28 days following the last dose of cabazitaxel OR have history of a vasectomy.
* Signed informed consent indicating an understanding of the purpose of the study and the necessary procedures and willingness to participate

Exclusion Criteria:

* History of severe hypersensitivity reaction (≥grade 3) to docetaxel and polysorbate 80 containing drugs
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments)
* Previous treatment with cabazitaxel
* Patients with Central Nervous System (CNS) metastasis. Patients without clinical signs or symptoms of CNS involvement are not required to have a CT/MRI of the brain
* Clinically significant cardiac disease within 6 months, including myocardial infarction, New York Heart Association (NYHA) Class III or IV heart disease, or left ventricular ejection fraction of < 50% at baseline for patients with a history of congestive heart failure.
* History of another malignancy in the previous 5 years with the exception of curatively treated non-melanomatous skin cancer.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness due to potential pharmacokinetic interactions of therapy with cabazitaxel.
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this trial.
* Unresolved toxicities from previous chemotherapy which has not resolved to ≤ grade 1 by CTCAE Version 4.02 criteria with the exception of alopecia or grade 2 peripheral neuropathy.
* Major surgery ≤ 2 weeks prior to the start of the study or who have not recovered from a previous surgery. (Placement of a venous access device within 2 weeks is permitted)

Min Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of patients progression-free survival after completion of treatment. | at end of treatment (up to 30 weeks)
  Treatment will continue until disease progression, intolerable side effects, or a maximum of 10 cycles of therapy. Progression-free survival defined as PSA progression, tumor progression in patients with measurable disease, or death.

SECONDARY OUTCOMES:
Number of patients that experience treatment-emergent adverse events | at end of each treatment cycle (up to 30 weeks)
  The assessment of safety will be based on the frequency and severity of adverse events. The incidence of treatment-emergent adverse events will be summarized by organ system, severity based on CTCAE (Common Terminology Criteria for Adverse Events) version 4.02, and relation to study drug by dose cohort. Adverse events assessed after each treatment cycle.
Number of patients with a prostate-specific antigen (PSA) response | at end of each treatment cycle (up to 30 weeks)
  PSA response defined as a 50% or more reduction in serum PSA concentration in patients with a serum PSA concentration of 20 μg/L or more at baseline and confirmed with a repeat PSA measurement after at least 3 weeks.
Change in geriatric assessments from baseline to end of therapy | every 2 cycles of therapy (6 weeks) up to 30 weeks
  Geriatric assessment to determine the relationship between functional ability or comorbidity and treatment response or toxicity. Patients will be have a geriatric assessment which will included a range of assessments, such as the Mini Mental Status Exam, Get Up and Go test, and the Geriatric Depression Scale, at baseline and after every 2 cycles of therapy.

OTHER OUTCOMES:
Change in circulating tumor cells (CTC) from baseline | at end of treatment (up to 30 weeks)
  Number of CTC at baseline and after treatment with cabazitaxel
Change in biomarkers from baseline | at 3 weeks (after one cycle)
  Level H2AX and M30 in CTCs at baseline and after treatment with cabazitaxel

CONTACTS AND LOCATIONS:
Overall Officials: Dale Shepard, Md, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center